CLINICAL TRIAL: NCT06177860
Title: Clinical Presentation, Coronary Angiographic Findings and Extent of Atherosclerotic Disease in Patients With Acute Coronary Syndrome Associated With Cocaine Use
Brief Title: Clinical and Atherosclerotic Characteristics of Patients With ACS Associated With Cocaine Use
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital El Cruce (Other)
Responsible Party: Principal Investigator, Maximiliano de Abreu, Principal Investigator, Hospital El Cruce
Other Study IDs: 00982023
Record Dates: First submitted 2023-11-29; First posted 2023-12-20 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Myocardial Infarction; Acute Coronary Syndrome; Cocaine Use; Cocaine Abuse
Keywords: Myocardial infarction; Acute Coronary Syndrome; Cocaine Use; Cocaine Abuse
MeSH Terms: conditions — Myocardial Infarction; Acute Coronary Syndrome; Cocaine-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cocaine use has increased in our country in recent decades. It is associated with cardiovascular events and early atherosclerotic disease. Acute coronary syndrome (ACS) is one of its most frequent and serious manifestations. There is a lack of scientific information on ACS associated with acute and chronic cocaine use in Argentina.

This study aims to describe the socioeconomic, clinical, and coronary angiographic characteristics, as well as the extent of atherosclerotic disease in patients with ACS associated with cocaine use, and to compare them with ACS not associated with cocaine use.

Methods: We propose an observational, analytical, single-center, two-phase study, with a retrospective and a prospective component. Patients with a diagnosis of ACS admitted to the coronary care unit of a high-complexity public hospital will be included. Clinical, biochemical, coronary angiographic, extracoronary atherosclerotic disease extension and prognostic variables will be described. These variables will be compared between patients with cocaine-associated ACS and non-cocaine-associated ACS.

DETAILED DESCRIPTION:
General objective:

- To identify socioeconomic, clinical, electrocardiographic, coronary angiographic, and atherosclerotic disease extent differences between ACS patients with a history of cocaine use and those without cocaine use.

Specific objectives:

To characterize and compare between both groups:

* Clinical characteristics.
* Coronary angiographic findings
* Extent of myocardial damage related and unrelated to ACS.
* Severe complications during hospitalization (mortality, resuscitated cardiac arrest, arrhythmias, use of IV inotropics and mechanical ventilatory support).
* Extent of noncoronary vascular disease.

Design:

A quantitative approach will be used, with an observational, analytical, single-center, two-stage design. In the retrospective stage, cases admitted from April 2019 to June 2023 for ACS will be included, based on data collected in the routine practice of the coronary care unit. In the prospective stage, all cases admitted to our institution for ACS from November 1, 2023, to November 2024 will be included.

Inclusion criteria:

* Age ≥18 years.
* Hospitalization with a diagnosis of ACS. For the prospective stage, acceptance to participate in the study and informed consent will be added.

Exclusion criteria:

Retrospective stage: patients who were not questioned about cocaine use. Prospective stage: patients who could not be interviewed to determine their history of cocaine use because of their clinical condition.

Procedures:

Two groups will be defined according to the history of cocaine use: cocaine-associated ACS and non-cocaine-associated ACS.

For the retrospective phase, all patients admitted to the coronary unit for ACS in the period established for the study will be reviewed. It is standard practice to ask about cardiovascular risk factors, history of substance use, including cocaine, and other clinical history. We expect to correctly identify cases of ACS associated and not associated with cocaine use.

In all cases included in both stages, the clinical, electrocardiographic, biochemical, and coronary angiographic characteristics and the extent of extra coronary atherosclerotic disease, complications, and prognosis will be described and compared between the two groups.

In the prospective phase of the study, where medically necessary, cardiac magnetic resonance imaging (MRI) will be performed to assess the extent of ACS-related and non-ACS-related myocardial necrosis and edema. Cardiac MRI findings will be compared between groups.

Clinical follow-up will be limited to hospitalization.

Main study variables and measurement instruments:

- ACS associated with cocaine and other substance use: They will be revealed by questioning, following evidence-based recommendations. ACS associated with cocaine use will be considered for those patients who verbally report the history.

* Clinical variables: Will be recorded on admission: age, weight and height, blood pressure, heart rate, cardiovascular risk factors (hypertension, diabetes, dyslipidemia, smoking), use of other substances (marijuana, using the same criteria as for cocaine), cardiovascular history (myocardial infarction, stroke, coronary revascularization, peripheral vascular disease, and heart failure).
* Electrocardiographic variables: 12-lead electrocardiograms will be performed on admission and during hospitalization to classify ACS as ST-elevation myocardial infarction (STEMI) or non-ST-elevation acute coronary syndrome (NSTEMI), to describe the location of ACS and to detect complications.
* Biochemical: a general and specific biochemical evaluation of ACS (CPK, CK mb, troponin, Pro BNP) will be performed. Peak enzymatic elevation of CPK and troponins will be used as a biochemical indicator of the extent of myocardial necrosis.
* Echocardiography: an assessment of ventricular function will be performed by measuring ejection fraction, diastolic dysfunction, and wall motility disorders. The presence of mechanical complications will be evaluated by this method.
* Extent and complexity of coronary atherosclerotic disease: coronary angiography will be used to define the extent and complexity of coronary lesions using the SYNTAX score. Also, an assessment of acute pathophysiological mechanisms related to ACS (thrombus, spasm, coronary dissection, as dichotomous variables: present or absent) will be performed.
* Extent of extra coronary atherosclerotic disease: ankle-brachial index (ABI) will be used as an indicator of peripheral vascular disease of the lower limbs. The presence, morphology, and extent of atherosclerotic plaque at the carotid level will be determined by carotid Doppler ultrasound.
* MRI: the degree of myocardial necrosis and edema related and unrelated to ACS will be assessed, as a manifestation of acute and chronic myocardial damage associated with ACS and cocaine use.

Statistical analysis:

Continuous variables will be described as mean and standard deviation in the case of normal distribution or median and interquartile range, and categorical variables will be described as numbers and percentages. Differences between groups for continuous variables will be evaluated with the T-test for variables with a normal distribution, and the Kruskal-Wallis test for nonparametric variables. Categorical variables will be compared using the chi-squared test and Fisher's exact test. Multiple logistic regression models will be developed to determine the independent association between cocaine use and the dependent variables of interest. Statistical analysis will be performed with the R Studio program.

Procedures to ensure the ethical aspects of the research:

All study procedures will be conducted following international ethical norms and standards to respect participant's rights and protect confidentiality.

In addition, all study procedures conform to the principles of the Declaration of Helsinki and CIOMS guidelines.

The research protocol was submitted for evaluation and approved by the Research Ethics Committee (REC) of the El Cruce Hospital.

For the retrospective stage, the research team will make every effort to contact patients who meet the inclusion criteria to request informed consent for their data to be analyzed, undertaking to guarantee the anonymity of personal data. For the prospective stage of the study, potentially eligible individuals will receive a detailed explanation of the objectives and procedures before enrollment. They will be asked to sign the informed consent form (ICF). Participation is voluntary and anonymity and confidentiality of information are compromised. At this stage, only cases that have signed the ICF will be included.

All information related to the study will be securely archived with access codes only available to the research team. Personal identification records will be kept separately from study records identified by code number. Data collection forms will be coded to maintain participant confidentiality. The local database will be protected with a password-protected access system. Study key codes linking participant identification numbers to other identifying information will be stored in a separate, locked file in a limited access area.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Hospitalization due to diagnosis of ACS, made by the treating medical team.

For the prospective stage, it will be added:

* Acceptance to participate in the study and willingness to sign the informed consent.

Exclusion Criteria:

* Patients who, due to their clinical condition, cannot be interviewed to determine their history of cocaine use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The biological sex and self-representation of gender identity of the patients will be recorded.
Study Population: Patients with acute coronary syndrome admitted to the coronary care unit of a high-complexity hospital.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Complexity and extent of coronary heart disease | During coronary angiography
  The Syntax Score (Synergy Between PCI With Taxus and Cardiac Surgery) will be quantified in patients with and without a history of cocaine use. A higher Syntax Score indicates a more complex coronary disease as well as worse prognosis. Score values of 0 to 22 are considered low complexity, 23 to 32 moderate complexity and >32 high complexity.
Clinical presentation as STEAMI, or NSTEAMI or unstable angina | Up to 24 hours of admission
  Differences between groups in clinical presentation as STEAMI, NSTEAMI or unstable angina will be based on the findings of the first electrocardiogram registred during admision, following the Fourth Universal Definition of Myocardial Infarction.
Mortality | During hospitalization (up to 30 days)
  Total mortality
Severe complications | During hospitalization (up to 30 days)
  A combined ouctome including: resuscitated cardiac arrest, complex arrhythmia requiring electrical cardioversion, use of inotropes, or mechanical ventilatory support.

SECONDARY OUTCOMES:
Extent of atherosclerotic vascular disease | During hospitalization (up to 30 days)
  The extent of extracoronary atherosclerotic vascular disease will be quantified by vascular Doppler of the carotids and lower limbs
Myocardial damage | During hospitalization (up to 30 days)
  The extent of ischemic and non-ischemic myocardial damage will be quantified by cardiac MRI.
Socioeconomic factors: unemployment | During hospitalization (up to 30 days)
  Unemployment (as a proportion) will be compared between patients with and without a history of cocaine use.
Socioeconomic factors: health insurance | During hospitalization (up to 30 days)
  Health insurance ownership (as a proportion) will be compared between patients with and without a history of cocaine use.
Socioeconomic factors: highest level of formal education | During hospitalization (up to 30 days)
  The highest level of formal education (as an ordinal variable from kindergarten = 1 to college = 8) will be compared between patients with and without a history of cocaine use.

CONTACTS AND LOCATIONS:
Overall Officials: Maximiliano de Abreu, PhD, Principal Investigator — Hospital El Cruce
Locations (1):
- Hospital El Cruce, San Juan Bautista, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided
It hasn't been decided yet

REFERENCES:
- [Result] Kim ST, Park T. Acute and Chronic Effects of Cocaine on Cardiovascular Health. Int J Mol Sci. 2019 Jan 29;20(3):584. doi: 10.3390/ijms20030584. PMID 30700023
- [Result] Lange RA, Hillis LD. Cardiovascular complications of cocaine use. N Engl J Med. 2001 Aug 2;345(5):351-8. doi: 10.1056/NEJM200108023450507. No abstract available. PMID 11484693
- [Result] Gatto L, Frati G, Biondi-Zoccai G, Versaci F. Cocaine and acute coronary syndromes: Novel management insights for this clinical conundrum. Int J Cardiol. 2018 Jun 1;260:16-17. doi: 10.1016/j.ijcard.2018.03.011. No abstract available. PMID 29622433
- [Result] Rezkalla SH, Kloner RA. Cocaine-induced acute myocardial infarction. Clin Med Res. 2007 Oct;5(3):172-6. doi: 10.3121/cmr.2007.759. PMID 18056026
- [Result] DeFilippis EM, Singh A, Divakaran S, Gupta A, Collins BL, Biery D, Qamar A, Fatima A, Ramsis M, Pipilas D, Rajabi R, Eng M, Hainer J, Klein J, Januzzi JL, Nasir K, Di Carli MF, Bhatt DL, Blankstein R. Cocaine and Marijuana Use Among Young Adults With Myocardial Infarction. J Am Coll Cardiol. 2018 Jun 5;71(22):2540-2551. doi: 10.1016/j.jacc.2018.02.047. Epub 2018 Mar 10. PMID 29535062
- [Result] Ma I, Genet T, Clementy N, Bisson A, Herbert J, Semaan C, Bouteau J, Angoulvant D, Ivanes F, Fauchier L. Outcomes in patients with acute myocardial infarction and history of illicit drug use: a French nationwide analysis. Eur Heart J Acute Cardiovasc Care. 2021 Dec 6;10(9):1027-1037. doi: 10.1093/ehjacc/zuab073. PMID 34453835
- [Result] Aquaro GD, Gabutti A, Meini M, Prontera C, Pasanisi E, Passino C, Emdin M, Lombardi M. Silent myocardial damage in cocaine addicts. Heart. 2011 Dec;97(24):2056-62. doi: 10.1136/hrt.2011.226977. Epub 2011 Jun 20. PMID 21690608
- [Result] US Preventive Services Task Force; Krist AH, Davidson KW, Mangione CM, Barry MJ, Cabana M, Caughey AB, Curry SJ, Donahue K, Doubeni CA, Epling JW Jr, Kubik M, Ogedegbe G, Pbert L, Silverstein M, Simon MA, Tseng CW, Wong JB. Screening for Unhealthy Drug Use: US Preventive Services Task Force Recommendation Statement. JAMA. 2020 Jun 9;323(22):2301-2309. doi: 10.1001/jama.2020.8020. PMID 32515821